CLINICAL TRIAL: NCT04367207
Title: African Covid-19 Critical Care Outcomes Study: An African, Multi-centre Evaluation of Patient Care and Clinical Outcomes for Patients With COVID-19 Admitted to High-care or Intensive Care Units
Brief Title: African Covid-19 Critical Care Outcomes Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Cape Town (Other)
Collaborators: University of KwaZulu (Other)
Responsible Party: Principal Investigator, Bruce Biccard, Professor, University of Cape Town
Other Study IDs: ACCCOS
Record Dates: First submitted 2020-04-27; First posted 2020-04-29 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Severe Acute Respiratory Syndrome Coronavirus 2
Keywords: Critical Care, Public Health

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients with COVID-19 referred to intensive care: Prospective observational cohort study of adult (≥18 years) patients referred to intensive care or high-care units in Africa with suspected or known COVID-19 infection in Africa

SUMMARY:
The infectious disease COVID-19, caused by coronavirus SARS-CoV-2 (severe acute respiratory syndrome coronavirus 2), has been declared a pandemic and an international healthcare emergency by the World Health Organization (WHO). It has spread across the globe, overwhelming healthcare systems by causing high rates of critical illness. Mortality from COVID-19 exceeds 4%, with older people with comorbidities being extremely vulnerable. It is expected that between 50-80% of the world's population may contract SARS-CoV-2 over the next two years. It is expected that the outcomes will be potentially worse in Africa, because firstly, there is a limited workforce, and secondly there are limited intensive care facilities and critical care resources across Africa to provide sufficient care. It is important therefore to establish what resources, comorbidities and interventions are potentially associated with either mortality or survival in patients with COVID-19 who are referred for critical care in Africa. Rapid dissemination of these findings may help mitigate mortality from COVID-19 in critical care patients in Africa. These points provide the rationale for the African COVID-19 Critical Care Outcomes Study (ACCCOS).

DETAILED DESCRIPTION:
The infectious disease COVID-19, caused by coronavirus SARS-CoV-2 (severe acute respiratory syndrome coronavirus 2), has been declared a pandemic and an international healthcare emergency by the World Health Organization (WHO). It has spread across the globe, overwhelming healthcare systems by causing high rates of critical illness. Mortality from COVID-19 exceeds 4%, with older people with comorbidities being extremely vulnerable.It is expected that between 50-80% of the world's population may contract SARS-CoV-2 over the next two years.

It is expected the outcomes to be potentially worse in Africa, because firstly, there is a limited workforce, and secondly there are limited intensive care facilities and critical care resources across Africa to provide sufficient care. It is estimated that there are 0.8 (95% confidence interval 0.3 to 1.45) critical care beds per 100,000 population in Africa. It is likely that the volume of unplanned admissions associated with COVID-19 will further adversely affect critical care outcomes in Africa,especially as the ability of healthcare systems in Africa to adapt and expand during the pandemic to meet the clinical workload is unknown. Furthermore, the patient outcomes in critical care is poorly documented in this under-resourced environment.

Most countries in Africa are still in the early phase of the epidemic which provides the opportunity to study the utilization of critical care resources and their impact on patient outcomes. It is important therefore to establish what resources, comorbidities and interventions are potentially associated with either mortality or survival in Africa. Rapid dissemination of these findings may help inform appropriate resource prioritisation and utilisation during the COVID-19 pandemic in Africa. These points provide the rationale for the African Covid-19 Critical Care Outcomes Study (ACCCOS).

Research questions

Primary outcome The primary outcome is in-hospital mortality in adult patients referred to intensive care or high-care units following suspected or known COVID-19 infection in Africa.

Secondary outcomes To determine the risk factors (resources, comorbidities and interventions) associated with mortality in adult patients with suspected or known COVID-19 infection in Africa.

The study is an African national multi-centre prospective observational cohort study of adult (≥18 years) patients referred to intensive care or high-care units in Africa with suspected or known COVID-19 infection in Africa. Patient follow up will be for a maximum of 30 days in-hospital.

This study will run between May to December 2020, with an interim analysis after 250 to 300 deaths registered in the study, or in June or July 2020 if this number of deaths has not been reported in the study. The reason for the interim analysis, is to potentially provide data which may be associated with improved outcomes in Africa, in timeous manner for possible implementation during this COVID-19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients at participating centres referred for high-care unit or intensive care unit admission who have suspected or known COVID-19

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (≥18 years) patients referred to intensive care or high-care units in Africa with suspected or known COVID-19 infection in Africa.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
In-hospital mortality | 8-12 months
  The primary outcome is in-hospital mortality in adult patients referred to intensive care or high-care units following suspected or known COVID-19 infection in Africa.

SECONDARY OUTCOMES:
Risk factors (resources, comorbidities and interventions) associated with mortality | 8-12 months
  To determine the risk factors (resources, comorbidities and interventions) associated with mortality in adult patients with suspected or known COVID-19 infection in Africa.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Biccard, Principal Investigator — University of Cape Town
Locations (1):
- Groote Schuur Hospital, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Biccard BM, Madiba TE, Kluyts HL, Munlemvo DM, Madzimbamuto FD, Basenero A, Gordon CS, Youssouf C, Rakotoarison SR, Gobin V, Samateh AL, Sani CM, Omigbodun AO, Amanor-Boadu SD, Tumukunde JT, Esterhuizen TM, Manach YL, Forget P, Elkhogia AM, Mehyaoui RM, Zoumeno E, Ndayisaba G, Ndasi H, Ndonga AKN, Ngumi ZWW, Patel UP, Ashebir DZ, Antwi-Kusi AAK, Mbwele B, Sama HD, Elfiky M, Fawzy MA, Pearse RM; African Surgical Outcomes Study (ASOS) investigators. Perioperative patient outcomes in the African Surgical Outcomes Study: a 7-day prospective observational cohort study. Lancet. 2018 Apr 21;391(10130):1589-1598. doi: 10.1016/S0140-6736(18)30001-1. Epub 2018 Jan 3. PMID 29306587
- [Background] Skinner DL, De Vasconcellos K, Wise R, Esterhuizen TM, Fourie C, Goolam Mahomed A, Gopalan PD, Joubert I, Kluyts HL, Mathivha LR, Mrara B, Pretorius JP, Richards G, Smith O, Spruyt MGL, Pearse RM, Madiba TE, Biccard BM, The South African Surgical Outcomes Study Sasos Investigators OBO. Critical care admission of South African (SA) surgical patients: Results of the SA Surgical Outcomes Study. S Afr Med J. 2017 Apr 25;107(5):411-419. doi: 10.7196/SAMJ.2017.v107i5.11455. PMID 28492122
- [Background] Pearse RM, Moreno RP, Bauer P, Pelosi P, Metnitz P, Spies C, Vallet B, Vincent JL, Hoeft A, Rhodes A; European Surgical Outcomes Study (EuSOS) group for the Trials groups of the European Society of Intensive Care Medicine and the European Society of Anaesthesiology. Mortality after surgery in Europe: a 7 day cohort study. Lancet. 2012 Sep 22;380(9847):1059-65. doi: 10.1016/S0140-6736(12)61148-9. PMID 22998715
- [Background] Biccard BM, Madiba TE; South African Surgical Outcomes Study Investigators. The South African Surgical Outcomes Study: A 7-day prospective observational cohort study. S Afr Med J. 2015 Jun;105(6):465-75. doi: 10.7196/samj.9435. PMID 26716164
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Peduzzi P, Concato J, Kemper E, Holford TR, Feinstein AR. A simulation study of the number of events per variable in logistic regression analysis. J Clin Epidemiol. 1996 Dec;49(12):1373-9. doi: 10.1016/s0895-4356(96)00236-3. PMID 8970487
- [Derived] African COVID-19 Critical Care Outcomes Study (ACCCOS) Investigators. Patient care and clinical outcomes for patients with COVID-19 infection admitted to African high-care or intensive care units (ACCCOS): a multicentre, prospective, observational cohort study. Lancet. 2021 May 22;397(10288):1885-1894. doi: 10.1016/S0140-6736(21)00441-4. PMID 34022988

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-08): https://cdn.clinicaltrials.gov/large-docs/07/NCT04367207/Prot_SAP_000.pdf